CLINICAL TRIAL: NCT00223366
Title: Studies on Normal and Inflamed Dental Pulp, NPY Regulation of Peripheral Human Nociceptors, Peripheral Mechanisms of Opioid Analgesia, Cannabinoid-induced Desensitization of TRPV1 Receptors Adrenergic Modulation of Trigeminal Nociceptors
Brief Title: In Vitro Studies on Pharmacological Regulation and Genetic Risk Factors of Peripheral Human Nociceptors
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair, Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20020071H; R01NS058655 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: Pain in teeth
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, sputum, oral mucosa tissue, teeth
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol is for a number of in vitro studies using human surgical biopsies and evaluating the pharmacology and genetics of human nociceptors ("pain detecting") neurons

DETAILED DESCRIPTION:
Purpose/Objectives

a. Specific Aims Specific Aim 1: Characterize in humans the effects of inflammation and neuronal degeneration on peripheral levels of NPY, and related Y receptors (Y1, Y2, Y5) in periradicular tissue.

Specific Aim 2: Determine whether NPY inhibits neurosecretion from peripheral terminals of capsaicin-sensitive neurons innervating normal versus inflamed tissue.

Specific Aim 3: Determine whether peripheral administration of NPY is analgesic and/or anti-allodynic in patients experiencing spontaneous pain and mechanical allodynia in a clinical model of inflammation with associated neuronal degeneration.

Specific Aim 4: Evaluate whether population characteristics are associated with altered pain reports. First, we will determine whether patients with the C1128 single nucleotide polymorphism (SNP) of the PreProNPY gene, whose phenotype confers substantially augmented peripheral NPY neurosecretion, report less pain compared with patients without this genetic polymorphism. Second, we will determine whether ethnic/cultural factors associated with an underserved minority population (Hispanics in the San Antonio area) are associated with altered pain reports.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate; identified indication to have a tooth extraction; 16-90 years old; diagnosis of normal pulp; or diagnosis of irreversible pulpitis requiring a symptom of spontaneous pain and positive and lingering response to pulp vitality test.

Exclusion Criteria:

* History of taking steroids within the last month; history of taking analgesics in the last four hours.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers between ages 16-90 y.o. presenting to the dental clinics within the University Health Science Center San Antonio for extraction of teeth.
Sampling Method: Non-Probability Sample
Enrollment: 2007 (Actual)
Dates: Start 2001-10 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
Effects of inflammation in periradicular tissues. | Immediately following tooth extraction and dental pulp procurement.
  Extracted human teeth are sectioned to obtain the crown dental pulp which is placed in a well plate. The pulp is moved every twenty minutes through proprietary substances for a total of 60 to 120 minutes depending on the specific experiment. After each 20 minute fraction, the buffer solution in each well plate is collected, labeled and placed in the -80 freezer along with the pulp sample.

SECONDARY OUTCOMES:
Altered pain reports. | 24 hour post-tooth extraction.
  Patients provide perceived pain within the first 24 hours post-extraction via a take-home pain postcard. The postcard has a Visual Analog Scale pain graft that the patient marks and returns via mail.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M. Hargreaves, DDS, PhD, Principal Investigator — University of Texas Health Science Center at San Antonio, Texas
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States